CLINICAL TRIAL: NCT02682108
Title: Diffusion-weighted Imaging Magnetic Resonance for Assessing Liver Fibrosis in Patients With Chronic Viral Hepatitis
Brief Title: Diffusion-weighted Imaging Magnetic Resonance for Assessing Liver Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Principle Investigator, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si237/2014
Record Dates: First submitted 2016-02-06; First posted 2016-02-15 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Fibrosis, Liver
Keywords: Hepatitis B; Hepatitis C; Fibrosis, Liver; Magnetic Resonance Imaging
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B; Hepatitis C | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diffusion-weighted imaging (Other): Magnetic resonance (MR) imaging examination of liver will be performed on a 3.0T Achieva MR scanner (Philips Medical Systems, The Netherlands). Diffusion-weighted imaging (DWI) will be performed using a single-shot echo-planar imaging during a single end expiratory breath-hold. A single observer placed circular regions of interest around 2.30 cm2 to measure mean signal intensity (SI) in the right hepatic lobe and the spleen for each b value, avoiding areas of artifact, vessels, and focal lesions. A monoexponential fit will be performed to calculate liver and spleen apparent diffusion coefficient (ADC) on the basis of ln(SI) as a function of b value, using all b values. Normalized liver ADC will be calculated as the ratio of liver ADC to spleen ADC.
  Interventions: Device: Diffusion-weighted magnetic resonance imaging (DW-MRI)

INTERVENTIONS:
Device: Diffusion-weighted magnetic resonance imaging (DW-MRI) — Magnetic resonance (MR) imaging examination of liver will be performed on a 3.0T Achieva MR scanner (Philips Medical Systems, The Netherlands). Diffusion-weighted imaging (DWI) will be performed using a single-shot echo-planar imaging during a single end expiratory breath-hold. A single observer placed circular regions of interest around 2.30 cm2 to measure mean signal intensity (SI) in the right hepatic lobe and the spleen for each b value, avoiding areas of artifact, vessels, and focal lesions. A monoexponential fit will be performed to calculate liver and spleen apparent diffusion coefficient (ADC) on the basis of ln(SI) as a function of b value, using all b values. Normalized liver ADC will be calculated as the ratio of liver ADC to spleen ADC.

SUMMARY:
Several noninvasive radiological techniques have been investigated for the diagnosis of liver fibrosis and cirrhosis among patients with chronic infection with hepatitis B virus or hepatitis C virus. Diffusion-weighted magnetic resonance imaging (DW-MRI) is a particularly appealing method for the diagnosis of liver fibrosis. The aims of this study are to evaluate the accuracy of DW-MRI in patients with chronic viral hepatitis for determining the stage of liver fibrosis.

DETAILED DESCRIPTION:
Among patients with chronic infection with hepatitis B virus or hepatitis C virus, evaluation of the stage of liver fibrosis is of major importance for determining prognosis and therapeutic decisions. Liver biopsy is a costly and invasive technique with associated mortality and morbidity. A typical biopsy fragment represents only 1/50,000 of the organ. Several noninvasive radiological techniques have been investigated for the diagnosis of liver fibrosis and cirrhosis. Diffusion-weighted magnetic resonance imaging (DW-MRI) is a particularly appealing method for the diagnosis of liver fibrosis. Because it is easy to implement, non-operator dependent, and process without the need for contrast agents. However, preliminary studies on small numbers of patients in which various hardware and sequencing profiles were used have reported inconsistent results for staging liver fibrosis with DW-MRI. The aims of this study are to evaluate correlation between stage of hepatic fibrosis and liver apparent diffusion coefficient (ADC) and normalized liver ADC with spleen assessed by DW-MRI in patients with chronic viral hepatitis B or C. Also, this study aim to evaluate factors that influence liver ADC and normalized liver ADC with spleen value for predicting the stage of liver fibrosis as well as to estimate the optimal cutoff values of DW-MRI for determining significant liver fibrosis (fibrosis stage ≥2) and advanced fibrosis (fibrosis stage ≥3).

ELIGIBILITY:
Inclusion Criteria:

* All naive patients with chronic hepatitis B or C infection who undergo liver biopsy examination for evaluating candidates for antiviral therapy will be invited to participate into this study

Exclusion Criteria:

* Other cause of chronic liver disease
* Contraindication for liver biopsy
* Contraindication for magnetic resonance imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The correlation coefficient of the stage of hepatic fibrosis and liver apparent diffusion coefficient as assessed by DW-MRI | At enrollment
  The primary aim of this study is to evaluate correlation between stage of hepatic fibrosis and liver apparent diffusion coefficient (ADC) and normalized liver ADC with spleen assessed by DW-MRI in patients with chronic viral hepatitis B or C.

SECONDARY OUTCOMES:
The optimal cutoff values of DW-MRI for determining the stage of liver fibrosis | At enrollment
  The aim of this study is to estimate the optimal cutoff values of DW-MRI for determining significant liver fibrosis (fibrosis stage ≥2) and advanced fibrosis (fibrosis stage ≥3).
The effects of hepatic steatosis, necroinflammation and hepatic iron on ADC values for determining the stage of liver fibrosis | At enrollment
  The aim of this study is to evaluate whether the degree of hepatic steatosis, necroinflammation, and hepatic iron affect the values of liver ADC and normalized liver ADC with spleen for determining the stage of liver fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make individual participant data available.

REFERENCES:
- [Background] Taouli B, Tolia AJ, Losada M, Babb JS, Chan ES, Bannan MA, Tobias H. Diffusion-weighted MRI for quantification of liver fibrosis: preliminary experience. AJR Am J Roentgenol. 2007 Oct;189(4):799-806. doi: 10.2214/AJR.07.2086. PMID 17885048
- [Background] Liaw YF, Kao JH, Piratvisuth T, Chan HL, Chien RN, Liu CJ, Gane E, Locarnini S, Lim SG, Han KH, Amarapurkar D, Cooksley G, Jafri W, Mohamed R, Hou JL, Chuang WL, Lesmana LA, Sollano JD, Suh DJ, Omata M. Erratum to: Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2012 update. Hepatol Int. 2012 Oct;6(4):809-10. doi: 10.1007/s12072-012-9386-z. No abstract available. PMID 26201529
- [Background] Soylu A, Kilickesmez O, Poturoglu S, Dolapcioglu C, Serez K, Sevindir I, Yasar N, Akyildiz M, Kumbasar B. Utility of diffusion-weighted MRI for assessing liver fibrosis in patients with chronic active hepatitis. Diagn Interv Radiol. 2010 Sep;16(3):204-8. doi: 10.4261/1305-3825.DIR.2810-09.1. Epub 2010 Jul 25. PMID 20658448
- [Background] Ferraioli G, Tinelli C, Dal Bello B, Zicchetti M, Lissandrin R, Filice G, Filice C, Above E, Barbarini G, Brunetti E, Calderon W, Di Gregorio M, Gulminetti R, Lanzarini P, Ludovisi S, Maiocchi L, Malfitano A, Michelone G, Minoli L, Mondelli M, Novati S, Patruno SF, Perretti A, Poma G, Sacchi P, Zanaboni D, Zaramella M. Performance of liver stiffness measurements by transient elastography in chronic hepatitis. World J Gastroenterol. 2013 Jan 7;19(1):49-56. doi: 10.3748/wjg.v19.i1.49. PMID 23326162
- [Background] Talwalkar JA, Kurtz DM, Schoenleber SJ, West CP, Montori VM. Ultrasound-based transient elastography for the detection of hepatic fibrosis: systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2007 Oct;5(10):1214-20. doi: 10.1016/j.cgh.2007.07.020. PMID 17916549
- [Background] Wang Y, Ganger DR, Levitsky J, Sternick LA, McCarthy RJ, Chen ZE, Fasanati CW, Bolster B, Shah S, Zuehlsdorff S, Omary RA, Ehman RL, Miller FH. Assessment of chronic hepatitis and fibrosis: comparison of MR elastography and diffusion-weighted imaging. AJR Am J Roentgenol. 2011 Mar;196(3):553-61. doi: 10.2214/AJR.10.4580. PMID 21343496
- [Background] Bonekamp S, Torbenson MS, Kamel IR. Diffusion-weighted magnetic resonance imaging for the staging of liver fibrosis. J Clin Gastroenterol. 2011 Nov-Dec;45(10):885-92. doi: 10.1097/MCG.0b013e318223bd2c. PMID 21716125
- [Background] Tosun M, Inan N, Sarisoy HT, Akansel G, Gumustas S, Gurbuz Y, Demirci A. Diagnostic performance of conventional diffusion weighted imaging and diffusion tensor imaging for the liver fibrosis and inflammation. Eur J Radiol. 2013 Feb;82(2):203-7. doi: 10.1016/j.ejrad.2012.09.009. Epub 2012 Nov 2. PMID 23122674
- [Background] Onur MR, Poyraz AK, Bozdag PG, Onder S, Aygun C. Diffusion weighted MRI in chronic viral hepatitis: correlation between ADC values and histopathological scores. Insights Imaging. 2013 Jun;4(3):339-45. doi: 10.1007/s13244-013-0252-x. Epub 2013 May 11. PMID 23666523